CLINICAL TRIAL: NCT05754411
Title: [14C] Study on Mass Balance and Biotransformation of STI-1558 in Healthy Chinese Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang ACEA Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPR-COV-103CN
Record Dates: First submitted 2023-02-03; First posted 2023-03-03 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]STI-1558 (Experimental)
  Interventions: Drug: [14C]STI-1558

INTERVENTIONS:
Drug: [14C]STI-1558 — Fasting oral administration of 600 mg [ 14C ] STI-1558 ( about 100 μCi ) solution.

SUMMARY:
This trial adopts a single-center, single-dose, single-period, non-randomized, open-label study design. It is planned to enroll 6~8 healthy male subjects, and each subject receives single oral administration of drug solution containing 600mg/approximately 100µCi [14C]STI-1558 under fasting conditions on trial D1. The whole blood, plasma, urine and stool samples are collected at specified time points/intervals during the trial. The pharmacokinetic parameters of the total radioactivity in plasma and whole blood, the material concentration ratios of the total radioactivity in plasma and whole blood, and the material balances are obtained by testing the total radioactivity of [14C]STI-1558 in plasma, whole blood, urine and feces. Meanwhile, using isotope tracer and mass spectrometry techniques, the main pathways and characteristics of metabolism and elimination of STI-1558 in humans are obtained through the quantification of radioactive metabolite profiles and the structure identification of the main metabolites in plasma, urine and feces of the subjects. The entire duration of trial is expected to be 5 months.

DETAILED DESCRIPTION:
The experiment was carried out in two steps :

Step 1 : Two qualified male subjects were enrolled in the study. After screening, the qualified subjects were admitted to the clinical research center after the D-2 was again verified by the inclusion and exclusion criteria. After admission, they were trained in medication, urine and feces collection procedures to ensure that they could perform relevant operations according to the program and SOP requirements. D-1 began to collect random urine samples ( -24 h~0 h ) and D-2 began to collect random fecal samples ( -48 h~0 h ). Subjects tested D1 morning fasting oral test drugs. All urine and feces samples excreted within the specified time interval of 0~336 h and blood samples at the specified time point of 0~168 h were collected. The test adopts the method of phased detection. According to the test results, it is judged whether the collection of blood, urine and feces samples can be terminated in advance or the collection needs to be continued. If the study finds that the collection time of biological samples exceeds the planned time ( i.e., blood 168 h, urine and feces 336 h ), the collection will be continued at an interval of 24 h ( or according to the researcher 's judgment, the integer multiple of 24 h ) until the judgment criteria for the termination of sample collection specified in the scheme are met. Safety monitoring continued until sample collection was completed.

Step 2 : 4-6 qualified male subjects were selected and blood, urine and feces samples were collected at the specified time points / intervals. The operation is the same as the first step. According to the test results of the first step test, determine whether the test process needs to be adjusted.

Criteria for terminating collection:

Excreta : The total radioactivity of biological samples ( urine + feces ) collected from each subject exceeded 90 % of the dose, and the total radioactivity of biological samples ( urine + feces ) collected for two consecutive days was less than 1 % of the dose ; radioactive blood samples : plasma radioactive concentration < 3 times plasma background value.

Finally, whether the subjects should terminate the collection of the corresponding samples was determined by the researchers based on the results of the radioactive test, the safety results and the actual situation, and the opinions of the sponsors.

All subjects were required to complete the test procedure according to the program requirements during their stay in the clinical research center. The subjects who met the radioactive recovery conditions were collected in the laboratory examination samples, and no clinically significant abnormalities were found in the clinical observation, and the group could be confirmed by the researchers. If the abnormality is found to have clinical significance, the subjects will need to remain in the research center for observation or after the comprehensive evaluation of the researchers, agree to leave the research center and return to the hospital for regular review ( according to the requirements of the researchers ), follow-up until the normal or abnormal level is returned to normal or not clinically significant or acceptable to the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign informed consent form;
* Chinese healthy male subjects between 18-45 years of age (inclusive);
* Weight: weight ≥ 50.0kg and body mass index (BMI) between 19.0~26.0kg/m2 (inclusive);
* Male subjects of childbearing potential who have no birth plans throughout the study period and for 12 months after the end of study, and agree to take contraceptive measures with their sexual partners during this period, such as condoms, contraceptive sponges, contraceptive gels, contraceptive films, intrauterine devices, oral or injected contraceptives (only suitable for the period after end of trial), subcutaneous implants (only suitable for the period after end of trial) or other contraceptive measures;
* Able to communicate well with the investigator and able to complete the trial in accordance with the protocol.

Exclusion Criteria:

Laboratory tests:

* Subjects who have clinically significant abnormalities through comprehensive physical examinations, vital signs, routine laboratory tests (blood routine, blood biochemistry, 4-item coagulation function, urine routine, stool routine + occult blood, etc.) and 12-lead ECG;
* Thyroid-stimulating hormone (TSH) > ULN (upper limit of normal); or free triiodothyronine (FT3) > ULN; or free thyroxine (FT4) > ULN;
* Blood amylase or lipase > ULN;
* Subjects who have any positive tests for hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, or combined HIV antigen/antibody test (primary screening);

Medication history:

* Subjects who have received any investigational products (including marketed products) or participated in any clinical trials with drugs/devices within 3 months prior to screening;
* Subjects who have used any drugs that inhibit or induce liver drug metabolizing enzymes within 30 days prior to screening (such as: inducers - barbiturates, carbamazepine, phenytoin, rifampicin, dexamethasone, rifabutin, rifapentine, etc.; inhibitors - SSRI antidepressants, cimetidine, diltiazem, macrolides, verapamil, imidazole antifungals, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines, etc.);
* Subjects who have taken any drugs that inhibit gastric acid secretion and gastric antiacids within 14 days prior to screening, such as H2 receptor antagonists (cimetidine, ranitidine, famotidine, nizatidine, roxatidine, etc.); proton pump inhibitors (omeprazole, lansoprazole, rabeprazole, pantoprazole, esomeprazole, etc.); and cholinergic receptor blockers (atropine, pirenzepine, etc.);
* Subjects who have used prescribed drugs, non-prescribed drugs, or health care medicines including western medicines or Chinese patent medicines within 30 days prior to administration (see exclusion criteria 6 and 7 for restrictions on liver drug metabolizing enzyme drugs, drugs that inhibit gastric acid secretion, and gastric antiacids); or have been vaccinated within 30 days prior to administration or plan to be vaccinated during the trial and within 30 days after end of trial;

Medical history and surgery history:

* Subjects with any history of clinically significant diseases or diseases or conditions that may affect the trial results in opinion of the investigator, including but not limited to history of motor system, nervous system, endocrine system, circulatory system, respiratory system, digestive system, urinary system and reproductive system diseases;
* Subjects with previous history of organic heart diseases (such as history of heart failure, history of myocardial infarction, history of angina pectoris), history of unexplained arrhythmia (such as history of ventricular tachycardia, history of QT prolongation syndrome) or symptoms or family history (with genetic evidences or close relatives who died suddenly from cardiac causes at a young age) of QT prolongation syndrome;
* Subjects with coagulation disorders, hemorrhagic diseases (such as hemophilia, purpura) or hemorrhagic symptoms (such as hematemesis, melena, hemorrhage of gastrointestinal tract, serious or recurrent epistaxis, hemoptysis, obvious hematuria or intracranial hemorrhage);
* Subjects who have suffered esophageal reflux or peptic ulcer diseases, or have received any previous surgical operations that may affect drug absorption (such as cholecystectomy) within 3 months prior to screening;
* Subjects who have received major surgeries within 6 months prior to screening or have surgical incisions that have not fully healed (see exclusion criteria 12 for surgical operation restrictions that may affect drug absorption); major surgeries include, but are not limited to, any surgeries with significant hemorrhage risks, prolonged general anesthesia periods, incisional biopsies or obvious traumatic injuries (except for appendicitis surgery or anal prolapse surgery that has recovered);
* Subjects with significant allergic conditions, including subjects who are clearly allergic to two or more other drugs or food ingredients; or subjects with previous history or family history of allergic skin diseases; or subjects who have special dietary requirements and cannot follow a unified diet;
* Subjects with mental disorders or previous history of mental disorders;
* Subjects with perianal diseases with concurrent hemorrhoids or regular/current hematochezia;
* Subjects with habitual constipation or diarrhea, irritable bowel syndrome, or inflammatory bowel diseases;

Living habits:

* Subjects who are alcoholics or regular drinkers within 6 months prior to screening, that is, consuming more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits with 40% alcohol or 150 mL of wine); or have positive results of alcohol breath tests during the screening period and baseline period; and cannot abstain during the trial;
* Subjects who smoke more than 5 cigarettes per day or habitually use nicotine-containing products in 3 months prior to screening, and cannot abstain during the trial;
* Subjects who abuse drugs or have used soft drugs (such as: marijuana) in 3 months prior to screening or hard drugs (e.g.: cocaine, amphetamines, phencyclidine, etc.) within 1 year prior to screening; or have positive results of urine drug abuse tests during the screening period and baseline period;
* Subjects who habitually drink grapefruit juice or excessive tea, coffee and/or caffeinated beverages and cannot abstain during the trial or have previous withdrawal syndrome;

Other:

* Subjects who cannot tolerate venipuncture, or have history of fear of needles and hemophobia;
* Subjects who are engaged in work with long-term exposure to radioactive conditions; or have significant radioactive exposure within 1 year prior to the trial (≥2 chest/abdominal CT, or ≥3 other types of X-ray examinations) or have participated in trials with radiolabeled drugs;
* Subjects who have had blood loss or donated more than 400 mL of blood within 3 months prior to screening, or received blood transfusion within 1 month;
* Subjects who have any other factors that are not suitable for participating in this trial in opinion of the investigator.
* Subjects who have any other factors that are not suitable for participating in this trial in opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Distribution Ratio of the Total Radioactivity in Whole Blood and in Plasma. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To investigate the distribution ratio of the total radioactivity in whole blood and plasma after oral administration of [14C]STI-1558 in healthy subjects。
Total Radioactivity in Whole Blood and in Plasma:AUC[0-t]. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To investigate the pharmacokinetic profiles of the total radioactivity in whole blood and plasma after oral administration of [14C]STI-1558 in healthy subjects.
Total Radioactivity in Whole Blood and in Plasma:Cmax . | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To investigate the pharmacokinetic profiles of the total radioactivity in whole blood and plasma after oral administration of [14C]STI-1558 in healthy subjects。
Total Radioactivity in Whole Blood and in Plasma:AUC[0-inf]. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration
  To investigate the pharmacokinetic profiles of the total radioactivity in whole blood and plasma after oral administration of [14C]STI-1558 in healthy subjects。
Total Radioactivity in Whole Blood and in Plasma:Tmax. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To investigate the pharmacokinetic profiles of the total radioactivity in whole blood and plasma after oral administration of [14C]STI-1558 in healthy subjects。
Total Radioactivity in Whole Blood and in Plasma:t1/2. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To investigate the pharmacokinetic profiles of the total radioactivity in whole blood and plasma after oral administration of [14C]STI-1558 in healthy subjects。
Total Radioactivity in the Excreta(Urine). | Urine samples collected:-24~0 hours before administration of [14C]STI-1558 and 0~8,8~24,24~48,48~72,72~96,96~120,120~144,144~168,168~192,192~216,216~240,240~264,264~288,288~312, 312~336 hours after administration.
  To perform the quantitative analysis of the total radioactivity in urine, and obtain the recovery of radioactivity and the main excretion pathways in humans after oral administration of [14C]STI-1558 in healthy subjects.
Total Radioactivity in the Excreta(Faeces). | Faeces samples collected:-48~0 hours before administration of [14C]STI-1558 and 0~24,24~48,48~72, 72~96,96~120,120~144,144~168,168~192,192~216, 216~240,240~264,264~288,288~312 ,312~336 hours after administration.
  To perform the quantitative analysis of the total radioactivity in faeces, and obtain the recovery of radioactivity and the main excretion pathways in humans after oral administration of [14C]STI-1558 in healthy subjects.

SECONDARY OUTCOMES:
Plasma Concentrations of STI-1558 (active compound AC1115):AUC[0-t]. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To perform the quantitative analysis of plasma concentrations of STI-1558 (active compound AC1115) using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) to evaluate the plasma pharmacokinetic parameters of STI-1558 (active compound AC1115).
Plasma Concentrations of STI-1558 (active compound AC1115):AUC[0-inf]. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To perform the quantitative analysis of plasma concentrations of STI-1558 (active compound AC1115) using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) to evaluate the plasma pharmacokinetic parameters of STI-1558 (active compound AC1115).
Plasma Concentrations of STI-1558 (active compound AC1115):Cmax. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To perform the quantitative analysis of plasma concentrations of STI-1558 (active compound AC1115) using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) to evaluate the plasma pharmacokinetic parameters of STI-1558 (active compound AC1115).
Plasma Concentrations of STI-1558 (active compound AC1115):Tmax . | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To perform the quantitative analysis of plasma concentrations of STI-1558 (active compound AC1115) using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) to evaluate the plasma pharmacokinetic parameters of STI-1558 (active compound AC1115).
Plasma Concentrations of STI-1558 (active compound AC1115):t1/2 . | TBlood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To perform the quantitative analysis of plasma concentrations of STI-1558 (active compound AC1115) using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) to evaluate the plasma pharmacokinetic parameters of STI-1558 (active compound AC1115).
Plasma Concentrations of metabolite M10:AUC[0-t]. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To perform the quantitative analysis of plasma concentrations of metabolite M10 using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) to evaluate the plasma pharmacokinetic parameters of metabolite M10.
Plasma Concentrations of metabolite M10:AUC[0-inf]. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To perform the quantitative analysis of plasma concentrations of metabolite M10 using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) to evaluate the plasma pharmacokinetic parameters of metabolite M10.
Plasma Concentrations of metabolite M10:Cmax. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To perform the quantitative analysis of plasma concentrations of metabolite M10 using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) to evaluate the plasma pharmacokinetic parameters of metabolite M10.
Plasma Concentrations ofmetabolite M10:Tmax . | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To perform the quantitative analysis of plasma concentrations of metabolite M10 using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) to evaluate the plasma pharmacokinetic parameters of metabolite M10.
Plasma Concentrations of metabolite M10:t1/2. | Blood samples collected:Within 1hour before administration of [14C]STI-1558 and 0.25、0.5、1、1.5、2、 3、4、6、8、12、24、48、72、120 、168 hours after administration.
  To perform the quantitative analysis of plasma concentrations of metabolite M10 using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) to evaluate the plasma pharmacokinetic parameters of metabolite M10.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | From administration of [14C]STI-1558 to Day14.
  To observe the safety of subjects after a single dose of [14C]STI-1558 until sample collection is complete.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Gaobo Boren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No